CLINICAL TRIAL: NCT00004209
Title: A Randomized Study of MVP 3 Versus 6 Cycles in Advanced Non-Small Cell Lung Cancer
Brief Title: Combination Chemotherapy in Treating Patients With Stage IIIB or Stage IV Non-small Cell Lung Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cancer Research UK (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: ICRF-95.240; CDR0000067457 (Registry Identifier: PDQ (Physician Data Query)); EU-99017
Record Dates: First submitted 2000-01-21; First posted 2004-09-16 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2007-06

CONDITIONS: Lung Cancer
Keywords: stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Cisplatin; Mitomycin; Vinblastine

INTERVENTIONS:
Drug: cisplatin
Drug: mitomycin C
Drug: vinblastine sulfate

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells. It is not yet known whether three courses of combination chemotherapy are more effective than six courses of combination chemotherapy for non-small cell lung cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of three courses of combination chemotherapy with that of six courses of combination chemotherapy in treating patients who have stage IIIB or stage IV non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the duration of symptom control, time to disease progression, survival, and quality of life in patients with stage IIIB or IV non-small cell lung cancer treated with 3 versus 6 courses of mitomycin, vinblastine, and cisplatin.

OUTLINE: This is a randomized, multicenter study. Patients are stratified by stage of disease (stage IIIB vs IV). Patients are randomized to 1 of 2 treatment arms: Arm I: Patients receive cisplatin IV over 4 hours, mitomycin IV, and vinblastine IV on day 1. Treatment repeats every 3 weeks for 3 courses in the absence of disease progression or unacceptable toxicity. Mitomycin is not administered during course 3. Arm II: Patients receive chemotherapy as in arm I. Treatment repeats every 3 weeks for 6 courses in the absence of disease progression or unacceptable toxicity. Mitomycin is not administered during courses 3 and 5. Quality of life is assessed after completion of 3 courses of chemotherapy for patients in arm I and after completion of 4, 5, and 6 courses for those in arm II. Patients may receive radiotherapy beginning after completion of chemotherapy.

PROJECTED ACCRUAL: A total of 310 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven stage IIIB or IV non-small cell lung cancer that is not eligible for surgery or radical radiotherapy

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Zubrod-WHO 0-2 Life expectancy: Not specified Hematopoietic: Hemoglobin greater than 10 g/dL WBC greater than 3,000/mm3 Platelet count greater than 100,000/mm3 Hepatic: Liver function tests no greater than 2 times normal (unless due to metastatic disease) Renal: Creatinine clearance greater than 60 mL/min EDTA clearance greater than 60 mL/min Other: No serious, uncontrolled, concurrent medical illness

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior conventional chemotherapy Endocrine therapy: Not specified Radiotherapy: See Disease Characteristics Surgery: See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1998-05

CONTACTS AND LOCATIONS:
Overall Officials: Ian E. Smith, MD, Study Chair — Royal Marsden NHS Foundation Trust
Locations (2):
- United Kingdom (2):
  - Royal Marsden NHS Trust, London, England
  - Aberdeen Royal Infirmary, Aberdeen, Scotland